CLINICAL TRIAL: NCT07035574
Title: Assessment of the Amount of Wear and Muscular Efficiency of 3D Printed Denture Teeth Versus Conventionally Fabricated Denture Teeth: A Cross-Over In Vivo Study
Brief Title: Assessment of Wear and Muscular Efficiency of 3D Printed Versus Conventional Denture Teeth: A Cross-Over In Vivo Study
Acronym: 3D-DENTURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, tuqa alazawy, Sponsor-Investigator, Principal Investigator, Prosthodontics Department, Faculty of Dentistry, Cairo University.", Cairo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TUQA2025DENTURE
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Edentulism
Keywords: 3D Printed Denture Teeth; Wear Analysis; Muscular Efficiency; Digital Dentistry

STUDY DESIGN:
Intervention Model Description: The study uses a crossover design where participants will receive two sets of complete dentures: one fabricated using conventional techniques and the other using 3D printing. This design minimizes individual variability and allows for direct comparison of outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Denture Teeth (Active Comparator): Participants will receive complete dentures fabricated using conventional techniques with prefabricated acrylic denture teeth.
  Interventions: Other: Conventional Denture Teeth
- 3D Printed Denture Teeth (Experimental): Participants will receive complete dentures fabricated using 3D printing technology with custom-designed denture teeth.
  Interventions: Other: 3D Printed Denture Teeth

INTERVENTIONS:
Other: Conventional Denture Teeth — Complete dentures fabricated using conventional techniques with prefabricated acrylic denture teeth.
  Arms: Conventional Denture Teeth
Other: 3D Printed Denture Teeth — Complete dentures fabricated using additive manufacturing techniques with advanced resin materials.
  Arms: 3D Printed Denture Teeth

SUMMARY:
This study aims to evaluate the wear resistance and muscular efficiency of denture teeth fabricated using two different methods: 3D printing and conventional techniques. The research is designed as a crossover in vivo study, where completely edentulous patients will receive both types of dentures sequentially. The primary outcome is the amount of wear observed in the denture teeth over time, while the secondary outcome is the muscular efficiency measured using electromyography (EMG). The study seeks to determine whether 3D printed denture teeth offer advantages in durability and functionality compared to conventionally fabricated denture teeth. Results from this study may provide valuable insights into improving the quality and comfort of dentures for edentulous patients.

DETAILED DESCRIPTION:
Complete dentures are a common treatment option for edentulous patients, providing essential functionality and aesthetics. With advancements in digital dentistry, 3D printing has emerged as a promising technique for fabricating denture teeth, offering potential benefits such as customization, faster production, and improved material properties. However, the long-term performance of 3D printed denture teeth compared to conventionally fabricated teeth remains under investigation.

This study is designed to assess two critical aspects of denture teeth performance: wear resistance and muscular efficiency. Wear resistance refers to the ability of denture teeth to withstand forces during chewing without significant degradation, while muscular efficiency evaluates how effectively the jaw muscles function with the dentures during activities like chewing and speaking.

The study will recruit completely edentulous patients aged 21-70 years from the Prosthodontics Department at Cairo University. Participants will receive two sets of complete dentures: one fabricated using conventional techniques and the other using 3D printing. The crossover design allows for direct comparison within the same group of patients, minimizing individual variability.

Primary impressions will be taken, followed by the fabrication of dentures using standardized protocols. The amount of wear will be measured by scanning the denture teeth at delivery and after three months of use. Muscular efficiency will be assessed using electromyography (EMG) to measure bite force at delivery and after three months.

This study is self-funded and conducted under the supervision of the Prosthodontics Department at Cairo University. Ethical approval has been obtained, and all participants will provide informed consent. The findings of this study are expected to contribute to the advancement of prosthodontic practices, offering evidence-based recommendations for the use of 3D printed denture teeth in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

Completely edentulous patients. Aged 21-70 years old. Able to read and sign the informed consent document. Class Ι maxilla-mandibular relationship. Free from temporomandibular disorders. Free from systemic diseases that could affect neuromuscular behaviors or muscular activities.

Edentulous condition falls within Class I and II cases based on the Prosthodontic Diagnostic Index (PDI) classification system for complete edentulism.

Exclusion Criteria:

Presence of major medical problems or severe chronic diseases. Poor residual ridge anatomy. Any intra-oral soft or hard tissue abnormalities. Flat, flabby, or knife-edge ridge anatomy.

-

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Amount of Wear | 6 months
  The amount of wear observed in denture teeth fabricated using conventional techniques versus 3D printing technology. Denture teeth will be scanned at delivery and after 3 months of use, and the wear will be quantified by comparing the scans.

SECONDARY OUTCOMES:
Muscular Efficiency | 6months
  Muscular efficiency will be assessed by measuring maximum bite force using electromyography (EMG) at delivery and after 3 months of use. The variation in bite force between conventional and 3D printed denture teeth will be analyzed.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to primary and secondary outcomes (amount of wear and muscular efficiency).
  Supporting documentation such as study protocol, statistical analysis plan, and informed consent form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available 6 months after study completion and will remain accessible for 5 years.
Access Criteria: Access will be granted to qualified researchers affiliated with academic institutions or research organizations.
  Researchers must submit a formal request and provide a detailed research proposal outlining the intended use of the data.
  Data will be shared via secure platforms or repositories, ensuring confidentiality and compliance with ethical guidelines.